CLINICAL TRIAL: NCT05854875
Title: RYGBP vs RYGBP With Fundus Resection for Morbid Obese Patients With Type 2 Diabetes. Evaluation of the Gastric Fundus in Glycemic Control. A Randomized Clinical Trial.
Brief Title: Diabetes Remission After RYGBP and RYGBP With Fundus Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Dimitrios Kehagias, Principal Investigator, University of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5378/35835
Record Dates: First submitted 2023-04-21; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Type 2 Diabetes; Morbid Obesity; Bariatric Surgery
Keywords: Gastric Fundus; Gastrointestinal Hormones
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RYGBP (Active Comparator): Laparoscopic Roux en Y Gastric Bypass
  Interventions: Procedure: Laparoscopic Roux en Y gastric bypass
- RYGBP + FR (Experimental): Laparoscopic Roux en Y Gastric Bypass with fundus resection
  Interventions: Procedure: Laparoscopic Roux en Y gastric bypass with fundus resection

INTERVENTIONS:
Procedure: Laparoscopic Roux en Y gastric bypass — Laparoscopic RYGBP included the creation of a small gastric pouch, with a 200cm biliopancreatic limb and a 150cm alimentary limb.
  Arms: RYGBP
Procedure: Laparoscopic Roux en Y gastric bypass with fundus resection — Laparoscopic RYGBP included the creation of a small gastric pouch, with a 200cm biliopancreatic limb and a 150cm alimentary limb. Fundus resection is further applied in this arm.
  Arms: RYGBP + FR

SUMMARY:
The goal of this randomized clinical trial is to evaluate glycemic control in patients with morbid obesity and type 2 diabetes after Roux-en-Y gastric bypass (RYGBP) and RYGBP with fundus resection. The main questions to answer are:

* Rate of diabetes remission and the role of the gastrointestinal hormones
* Whether fundus resection leads to improved glycemic control

Patients will randomly undergo typical RYGBP or RYGBP with fundus resection. Gastrointestinal hormones profile [ghrelin, glucagon-like peptide-1 (GLP-1), peptide YY (PYY), glucagon], glucose levels and insulin response will be measured preoperatively, at 6 months and at 12 months, during 120-min OGTT.

ELIGIBILITY:
Inclusion Criteria:

* morbid obesity (ΒΜΙ ≥ 40)
* type II diabetes mellitus (T2DM)
* duration of T2DM shorter than 8 years

Exclusion Criteria:

* pregnancy
* type 1 diabetes
* previous gastrointestinal surgeries
* alcohol consumption
* depression
* no compliance

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-22 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Diabetes remission in both groups | At 6 months and 12 months postoperatively
  Change in HbA1c levels
Change in fasting and postprandial glucose levels | At 6 months and 12 months postoperatively
  Glucose levels (mg/dl)
Change in insulin levels, fasting and postprandial | At 6 months and 12 months postoperatively
  Insulin levels (μIU/ml)
Change in HOMA - IR | At 6 months and 12 months postoperatively
  HOMA IR calculation with glucose (mg/dl) and insulin (mU/L)
Change in ghrelin levels | At 6 months and 12 months postoperatively
  Fasting and postprandial ghrelin levels (pg/ml)
Change in GLP-1 levels | At 6 months and 12 months postoperatively
  Fasting and postprandial GLP-1 levels (pg/ml)
Change in PYY levels | At 6 months and 12 months postoperatively
  Fasting and postprandial PYY levels (ng/ml)
Change in glucagon levels | At 6 months and 12 months postoperatively
  Fasting and postprandial glucagon levels (pg/ml)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Patras, University Hospital of Patras, Pátrai, Rio, Greece

IPD SHARING:
Plan to Share IPD: No